CLINICAL TRIAL: NCT07127315
Title: A Prospective Study Assessing Gonadotropin-Releasing Hormone Agonists Benefit in Preserving the Ovarian Function in Premenopausal Breast Cancer Patients During Chemotherapy
Brief Title: Assessing Gonadotropin-Releasing Hormone Agonists Benefit in Preserving the Ovarian Function in Premenopausal Breast Cancer Patients During Chemotherapy
Status: Completed | Type: Observational
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Fatma Mohsen Kamal, Assistant Lecturer of Clinical Oncology, Faculty of Medicine, Helwan University, Helwan, Egypt., Helwan University
Other Study IDs: 51-2022
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Gonadotropin Releasing Hormone Agonists; Ovarian Function; Premenopausal; Breast Cancer; Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Gonadotropin-Releasing Hormone; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Patients received chemotherapy plus a gonadotropin-releasing hormone agonist.
  Interventions: Drug: Gonadotropin-releasing hormone agonist
- Control group: Patients received chemotherapy alone.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Gonadotropin-releasing hormone agonist — Patients received chemotherapy plus a gonadotropin-releasing hormone agonist.
  Groups: Intervention group
Drug: Chemotherapy — Patients received chemotherapy alone.
  Groups: Control group

SUMMARY:
The purpose of this study is to investigate the benefits of gonadotropin-releasing hormone agonist administration during chemotherapy on preserving ovarian function and Fertility in Premenopausal breast cancer patients, as assessed by anti-mullerian hormone levels, luteinizing hormone (LH), follicle-stimulating hormone (FSH), and estradiol (E2) levels.

DETAILED DESCRIPTION:
The annually estimated number of females diagnosed with cancer is about 6.6 million, 10% of whom are premenopausal.

To minimize the risk of ovarian dysfunction and infertility for these patients, ovarian reserve differs widely from one female to another, but it could be assessed by Ultrasound to reveal antral follicle count (AFC). Also, the hormonal levels of anti-Müllerian hormone (AMH), estradiol (E2), and follicle-stimulating hormone FSH are valuable indicators for fertility.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal female patients 18-45 years.
* Female patients with pathologically confirmed breast cancer and receiving a chemotherapy regimen, either adjuvant or neoadjuvant, containing a gonadotoxic agent.
* Female patients with performance status (PS) ≤ 2.

Exclusion Criteria:

* All female Patients with metastatic cancer.
* Patients underwent total abdominal hysterectomy and bilateral salpingo-oophorectomy, or patients received radiotherapy on the pelvis.
* Patient with end-organ failure.
* Patients with performance status >2.
* Male with breast cancer.
* Post-menopausal females.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Premenopausal female patients
Study Population: 100 females with early-stage breast cancer were recruited from the Clinical Oncology Department at Helwan University Hospital for this interventional prospective cross-sectional case-control cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Anti-mullerian hormone level | Immediately post-procedure (Up to 1 hour)
  Anti-mullerian hormone level was calculated.

SECONDARY OUTCOMES:
Follicle-stimulating hormone level | Immediately post-procedure (Up to 1 hour)
  Follicle-stimulating hormone level was calculated.
Estradiol level | Immediately post-procedure (Up to 1 hour)
  Estradiol (E2) level was calculated.
Disease-free survival | 2 years post-procedure
  Disease-free survival (DFS) was calculated.
Overall survival | 2 years post-procedure
  Overall survival (OS) was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Helwan University, Helwan, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.